CLINICAL TRIAL: NCT01133054
Title: Physiologic Evaluation of Anomalous Right Coronary Artery Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Associate professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-0908-010-060
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Vessel Anomalies
Keywords: Coronary Vessel Anomalies
MeSH Terms: conditions — Coronary Vessel Anomalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low FFR (Experimental): FFR<0.75
  Interventions: Procedure: revascularization
- high FFR (No Intervention): FFR > 0.75

INTERVENTIONS:
Procedure: revascularization — surgery or stenting
  Other Names: other names are not available
  Arms: low FFR

SUMMARY:
The anomalous origin of right coronary artery (RCA) is a rare coronary anomaly. Recently, the detection of this anomaly has been more frequent as the use of cardiac multidetector computed tomography has become more popular. It can cause myocardial ischemia, syncope and sudden cardiac death. Surgical repair is generally recommended for symptomatic patients. However, there is controversy concerning the proper evaluation and treatment strategy for patients without documented myocardial ischemia.

The stenotic lesion of anomalous origin of RCA will be assessed by fractional flow reserve (FFR).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as anomalous origin of right coronary artery from left coronary cusp

Exclusion Criteria:

* poor compliance
* need for percutaneous coronary intervention to significant coronary lesion
* failure of FFR for anomalous origin of right coronary artery

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cardiac death | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon KOO, M.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea